CLINICAL TRIAL: NCT03204838
Title: STUDY TITLE IDH1/IDH2 Mutation Frequency in Acute Myeloblastic Patients and Myelodysplasticsyndromes, Clinical Response to Treatment
Brief Title: IDH1/IDH2 Mutation Frequency in Acute Myeloblastic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, ADOLFO MARTINEZ TOVAR, Principal Investigator, Hospital General de México Dr. Eduardo Liceaga
Other Study IDs: Hospital General de Mexico
Record Dates: First submitted 2017-06-25; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: IDH1, IDH2, MUTATION, AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Retrospective phase clinical and molecular data of patients without treatment with morphological, genetic, immunophenotype classification. Molecular biology (AML-ETO, PMR-RAR alpha, Inv 16, FLT 3, CEBP mutation 50 cases , 100 controls. Address Hospital General de Mexico , Hematology service ( external consult and transfusional area). (Lysis Buffer)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AML patients: Adult AML patients with the IDH mutation test performed at diagnosis.
  Interventions: Genetic: IDH mutation test performed at diagnosis

INTERVENTIONS:
Genetic: IDH mutation test performed at diagnosis — Observation of the test result

SUMMARY:
This leukemia is characterized by a poor prognosis for most patients, as they have a high relapse rate despite aggressive treatment with chemotherapy agents and allogeneic bone marrow transplantation. It has been proposed that relapse can be attributed to a leukemic cells population with quiescence properties that are resistant to chemotherapy, known as leukemic stem cells (LSCs). Clinical trials shown a major LSCs percentage than diagnosis correlated with worst prognosis or minimal residual disease with AML.

AML is most common in adults and represents about 40% of all leukemia types in American Continent. In Mexican patients with AML age median is 32 years, lower than other international series. Genomic and functional studies have identified two classes of mutations, which cooperate during AML development.

Somatic mutations have been identified recently that codify for isocitrate dehydrogenase (IDH). These genes codify key metabolic enzymes, which convert isocitrate into α-ketoglutarate (α-KG).15-16From which IDH1 and IDH2 genes presenta high frequency of mutations in AML and other types of tumors. IDH mutations affect mainly active site residues (for example, IDH1 R132, IDH2 R140 or IDH2 R172), resulting in the normal enzymatic function loss abnormally converting α-KG to 2-hydroxiglutarate (2-HG).

"Oncometabolyte" 2-HG may competitively inhibit multiple α-KG depending dioxygenases, including key epigenetic regulators as histones demethylases and TET proteins. Consequently, IDH mutations are associated with chromatin alterations including global alteration of histones and NDA methylation. This is the reason of the need to identify such mutations of genes (IDH1/IDH2) in patients with SMD and AML entering Hematology service of the Hospital General de Mexico from 2017 to 2019, and determine clinical impact in prognosis and monitoring the response to therapy, as well as prognosis and survival.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a heterogeneous cancer implying accumulation of mature cells. This leukemia is characterized by a poor prognosis for most patients, as they have a high relapse rate despite aggressive treatment with chemotherapy agents and allogeneic bone marrow transplantation. It has been proposed that relapse can be attributed to a leukemic cells population with quiescence properties that are resistant to chemotherapy, known as leukemic stem cells (LSCs). Clinical trials shown a major LSCs percentage than diagnosis correlated with worst prognosis or minimal residual disease with AML.

AML is most common in adults and represents about 40% of all leukemia types in American Continent. In Mexican patients with AML age median is 32 years, lower than other international series.

AML may be classified in 8 sub-types based on FAB Classification (French-American-British Classification). FAB Classification is based on morphology and cytogenetic. Sub-types are M0 to M7, based on the type of leukemia cells and their maturity. Other classification system used is the one of the World Health Organization (WHO) that classifies the types of leukemia based on genetic/molecular alteration or existence of other potential factors impacting clinical prognosis. The Hospital General de Mexico classifies the leukemia types based on morphologic, immunophenotype, genetic and sometimes in molecular criteria.

Genomic and functional studies have identified two classes of mutations, which cooperate during AML development. Class I mutations, which confer proliferative and survival advantage to hematopoietic stem cells, an example is the occurrence of mutations in NRAS or KRAS genes, or mutations affecting receptor tyrosine kinase FLT3.Class II mutations characterize for promoting self-renewal and blocking differentiation of hematopoietic stem cells. These mutations include certain translocation, an example of this type of mutations is gene MLL1 derived from t(8;21) (AML1-ETO).Major mutations in AML are commonly detected in cytogenetically Normal (CN) cases representing 40% to 50% of all AML.

Such aberrations have demonstrated impacting prognosis of patients with AML. These genes include: FLT3, NPM1, CEBPA, MLL, NRAS, KIT, WT1, RUNX1, TET2, IDH1/2, DNMT3A, ASXL1, PHF6. For example, mutations in FLT3 (37%-46% of patients) indicate poor prognosis. On the contrary, mutations in NPM1 (48%-53% of patients) and CEBPA (13% to 15% of patients) indicate a better prognosis. AMLis a neoplastic clonal disease that originates from progressive accumulation of genetic and epigenetic aberrations affecting mechanisms regulating proliferation and differentiation of hematopoietic trunk cells (HTC). However, impact of these mutations in survival and chemo resistance to new therapeutic agents in LSCs, including emergent therapies against LSCs, which have not been described. In the Hospital General de Mexico, the prognosis of LAM at 5 years is only 30%. For this, it is necessary to detect mutation pattern of genes that may contribute to AML development or prognosis in Mexican patients of the Hospital General de México.

Somatic mutations have been identified recently that codify for isocitrate dehydrogenase (IDH). These genes codify key metabolic enzymes, which convert isocitrate into α-ketoglutarate (α-KG).15-16From which IDH1 and IDH2 genes presenta high frequency of mutations in AML and other types of tumors. IDH mutations affect mainly active site residues (for example, IDH1 R132, IDH2 R140 or IDH2 R172), resulting in the normal enzymatic function loss abnormally converting α-KG to 2-hydroxiglutarate (2-HG).

"Oncometabolyte" 2-HG may competitively inhibit multiple α-KG depending dioxygenases, including key epigenetic regulators as histones demethylases and TET proteins. Consequently, IDH mutations are associated with chromatin alterations including global alteration of histones and NDA methylation. This is the reason of the need to identify such mutations of genes (IDH1/IDH2) in patients with SMD and AML entering Hematology service of the Hospital General de Mexico from 2017 to 2019, and determine clinical impact in prognosis and monitoring the response to therapy, as well as prognosis and survival..

ELIGIBILITY:
Inclusion Criteria:

Signed written informed consent according to ICH/GCP and national local laws

AML patients; >18 years IDH mutation test perfomed at diagnosis

Exclusion Criteria:

Patients whom don't continue treatment. AML-M3 subtype according to the FAB

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AML patients without treatment with morphological, genetic, immunophenotype classification.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-10 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-05 (Estimated)

PRIMARY OUTCOMES:
Identify the mutation frequency of IDH1/IDH2 genes in patients with AML entering Hematology service of the HGM and clinical impact in treatment respons | At two years from study entry
  Number of patients with the IDH mutation in AML at initial diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: ADOLFO A Martinez Tovar, phD, Principal Investigator — Hospital General de Mexico
Locations (1):
- Ciudad de Mexico, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gutierrez-Malacatt H, Ayala-Sanchez M, Aquino-Ortega X, Dominguez-Rodriguez J, Martinez-Tovar A, Olarte-Carrillo I, Martinez-Hernandez A, C CC, Orozco L, Cordova EJ. The rs61764370 Functional Variant in the KRAS Oncogene is Associated with Chronic Myeloid Leukemia Risk in Women. Asian Pac J Cancer Prev. 2016;17(4):2265-70. doi: 10.7314/apjcp.2016.17.4.2265. PMID 27221928
- [Result] Alonso-Rangel L, Benitez-Guerrero T, Martinez-Vieyra I, Cisneros B, Martinez-Tovar A, Winder SJ, Cerecedo D. A role for dystroglycan in the pathophysiology of acute leukemic cells. Life Sci. 2017 Aug 1;182:1-9. doi: 10.1016/j.lfs.2017.06.004. Epub 2017 Jun 4. PMID 28591567
- [Result] Santoyo-Sanchez A, Ramos-Penafiel CO, Saavedra-Gonzalez A, Gonzalez-Almanza L, Martinez-Tovar A, Olarte-Carrillo I, Collazo-Jaloma J. [The age and sex frequencies of patients with leukemia seen in two reference centers in the metropolitan area of Mexico City]. Gac Med Mex. 2017 Jan-Feb;153(1):44-48. Spanish. PMID 28128805
- [Result] Olarte Carrillo I, Ramos Penafiel C, Miranda Peralta E, Rozen Fuller E, Kassack Ipina JJ, Centeno Cruz F, Garrido Guerrero E, Collazo Jaloma J, Nacho Vargas K, Martinez Tovar A. Clinical significance of the ABCB1 and ABCG2 gene expression levels in acute lymphoblastic leukemia. Hematology. 2017 Jun;22(5):286-291. doi: 10.1080/10245332.2016.1265780. Epub 2016 Dec 14. PMID 27960630